CLINICAL TRIAL: NCT02415907
Title: Interventional, Open-label, Two Single Dose, Fixed-sequence Study Investigating the Absorption, Metabolism and Excretion (AME) of Idalopirdine Following a Single Oral Dose of Lu AF67708 ([Ethyl-1-14C]-Idalopirdine) and Lu AF67709 ([Benzyl-7-14C]-Idalopirdine) in Healthy Men
Brief Title: Investigating the Absorption, Metabolism and Excretion (AME) of Idalopirdine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15836A; 2013-004001-28 (EudraCT Number)
Record Dates: First submitted 2015-04-07; First posted 2015-04-14 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Idalopirdine (Experimental): Period I: Initial administration of Lu AF67709 single dose at baseline.
  Period II: Administration of Lu AF67708 single dose (week 4)
  Interventions: Drug: [ethyl-1-14C]-idalopirdine; Drug: [benzyl-7-14C]-idalopirdine

INTERVENTIONS:
Drug: [ethyl-1-14C]-idalopirdine — 120 mg/2.40 MBq Lu AF67708 ([ethyl-1-14C]-idalopirdine) in one capsule for oral administration, single dose
  Other Names: Lu AF67708
Drug: [benzyl-7-14C]-idalopirdine — 120 mg/2.40 MBq Lu AF67709 ([benzyl-7-14C]-idalopirdine) in one capsule for oral administration, single dose
  Other Names: Lu AF67709

SUMMARY:
The purpose of this study is to investigating the absorption, metabolism and excretion of radio labelled single doses of idalopirdine in healthy men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* aged between 40-60 years (inclusive)
* BMI in the range 19 and 30 kg/m2 (minimum weight 60 kg)

Exclusion Criteria:

* The subject has previously been dosed with idalopirdine.

Other protocol defined inclusion and exclusion criteria do apply

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Cumulative amounts of radioactivity excreted in urine and faeces (% of dose) | 0 to 168 hours
Pharmacokinetic (PK) of idalopirdine and radioactivity in plasma (Cmax, tmax, AUC, t1/2, oral clearance and apparant volume of distribution. (composite outcome measure) | 0 to 168 hours
  PK parameter:

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck, Study Director — LuncbeckClinicalTrials@Lundbeck.com
Locations (1):
- GB802, Leeds, United Kingdom